# **Protocol**

SPREAD-NET: PRactices Enabling Adapting and Disseminating in the Safety NET

NCT02325531

6/2/2016

#### **INSTRUCTIONS:**

- **All sections are required**. If a section does not apply to your project please enter "N/A." The level of detail required for each section will vary with the complexity of your project.
- If your study has multiple aims, break each section down to address each aim of the study, as appropriate.
- Delete all instructions (italics).
- See the <u>Research Compliance</u> website for guidance and information on a number of topics including vulnerable populations, consent, inclusion of non-English speakers, genetic research, and data sharing.
- If you are doing a data-only study with no prospective or interventional components, use the **Data Only Protocol Template** instead.

#### 1. Protocol Title

SPREAD-NET: Practices Enabling Implementation and Adaptation in the Safety Net

# 2. Objectives

We propose to compare the effectiveness of different 'support strategies' at helping diverse community health clinics (CHCs) sustainably implement an intervention shown to reduce patients' cardiovascular disease (CVD) event risk. Kaiser Permanente developed and implemented the 'ALL Initiative' (a.k.a. 'ALL'), a clinic-level intervention designed to increase rates of adult patients with diabetes mellitus (DM) or CVD who are prescribed cardio-protective medications (statins and ACE-Inhibitors) according to evidence-based guidelines. After ALL was shown to be highly effective in Kaiser Permanente's integrated care setting, our team demonstrated the feasibility of adapting it for successful implementation in 11 CHCs - with the help of substantial implementation support. The next step in this body of research is to identify the amount and type of support needed to effectively implement and sustain this intervention in a greater number of CHCs. To that end, we will conduct a trial in which 30 CHCs are clusterrandomized to receive low, medium, or high-intensity support in implementing ALL. We will conduct this work with CHC members of OCHIN, a community health information technology network that hosts one of the nation's largest CHC electronic health record (EHR) platforms; study CHCs share a single, linked EHR. Guided by the Practice Change Model and RE-AIM framework, we will use mixed-methods to:

Aim 1: Compare how effectively the low, medium, and high-intensity strategies support the CHCs' implementation of ALL, and assess change in rates of clinic patients with (i) guideline-appropriate cardioprotective prescriptions, and (ii) controlled blood pressure and low-density lipoprotein, as associated with implementation supported by the different strategies;

Aim 2: Assess the strategies' effectiveness at supporting intervention sustainability over 3 years; and

Aim 3: Identify clinic characteristics associated with success at different levels of support. Our team includes CHC clinicians, and experts in dissemination and implementation (D&I), health economics, and health services research mixed-methods. Our study is designed to inform future implementation of ALL as well as other interventions known to improve outcomes among CHC patients with DM / CVD. Our results could also have high impact on D&I science, by comparing practical, generalizable methods for supporting the implementation of clinical innovations in CHCs and other ambulatory settings.

Research questions: What are the characteristics of clinics that achieve sustained change even with less implementation support, and of those that do not achieve change even with more support?

# 3. Background

A major barrier to the timely dissemination of evidence-based interventions is a lack of knowledge about efficient, replicable strategies for supporting the implementation of tested interventions in routine care. This is particularly relevant to intervention implementation in safety net Community Health Centers (CHCs\*).<sup>1-16</sup>

Disseminating successful interventions in diverse primary care settings could significantly improve the health of patients with DM / CVD nationwide. Yet few studies have focused on comparing effective strategies for supporting change in health care settings. <sup>5,79-91</sup> Thus an important barrier to the widespread dissemination of evidence-based interventions such as ALL is a lack of knowledge about the most effective strategies for supporting sustainable implementation in diverse care settings. <sup>1,3,5,8-11,15,21,22,24,42,44,79-88,92-97</sup> This limitation is particularly problematic for the Community Health Centers (CHCs) in our health care 'safety net', <sup>1,13,14</sup> which care for millions of underserved patients, and are expected to serve millions more through the Affordable Care Act. <sup>98-100</sup> Rapid, effective implementation of interventions shown to improve care delivery and health outcomes could ensure that CHC patients benefit from cutting-edge clinical knowledge. Although the need is well-acknowledged, we know of no previous randomized trial comparing strategies for supporting consistent, reliable implementation of evidence-based care in CHCs. <sup>7,10,12,101</sup>

This study will address the lack of knowledge about effective implementation support strategies. We propose to compare the effectiveness of 3 replicable strategies for supporting the implementation of the ALL Initiative in CHCs. These strategies have been shown to be effective and feasible in CHCs. We will conduct a pragmatic trial in which 30 CHCs are cluster-randomized to receive low, medium, or high-intensity implementation support.

We propose to address an important barrier to such dissemination - the lack of knowledge about the most effective strategies for supporting CHCs' implementation of evidence-based interventions. 1,13,14,45,79-91,93 This work is positioned to have broad impact. Understanding how to efficiently support implementing the evidence-based ALL Initiative in CHCs could reduce CVD event risk in patients with CVD / DM nationwide, improving health outcomes and reducing care costs. While this project focuses on ALL in CHCs, we will discover generalizable strategies for implementing ALL in other primary care settings and also for supporting CHCs' implementation of other interventions shown to improve CVD /DM outcomes, and other morbidities.

#### 4. Study Design

We will conduct a cluster-randomized, prospective, pragmatic trial with 3 arms (Figure 3). In months 1-18, we will collect baseline data via a survey of all study sites, and refine the toolkit. At the start of Implementation Year 1 (study month 19), 30 CHCs will be randomized to receive low, medium, or high-intensity support in implementing the ALL Initiative. Guided by RE-AIM and the Practice Change Model, we will use mixed methods to assess how effectively the different levels of intensity support intervention uptake, guideline-based prescribing, and patient health (Aim 1), and sustainability over 3 years (Aim 2). We will identify clinic-level factors associated with each support strategy's effectiveness and sustainability (Aim 3), and adapt as possible. We will also conduct a cost analysis.

Arm 1 ('Low' intensity support) components: TOOLKIT. The point person will receive the implementation toolkit (paper and electronic form) at the start of Implementation Year 1. Toolkit components are ready for

use except as noted. EHR-based tools, built in OCHIN's EHR, will be activated at that time. The toolkit will include annual 1-hour 'Basic Webinars' open to the study point person, and hosted by the research team.

Arm 2 ('Medium' intensity support) components: Arm 2 CHCs will receive the TOOLKIT as above. TRAIN-THE-TRAINER: The study 'point person' will receive extensive implementation training at a 2-day in-person meeting in Portland, OR. Our implementation specialists will teach participants how to use the ALL toolkit and how to train others to use it. Training content will include necessary elements as identified by (i) our previous research, (ii) the baseline survey), (iii) the study team and the SPREAD-NET advisory group. Trainees will be asked to train staff at their clinic within 6 weeks after the in-person event. ADAPTIVE WEBINARS: The point people will join quarterly 1-hour webinars hosted by the research team. One webinar will include the content from the Toolkit's 'Basic' webinars. The other three will include content to reinforce and augment information from the in-person training, and to address factors that the Practice Change Model identifies as influential on intervention implementation in primary care settings. These webinars will provide a forum for group discussion and best practice sharing. We will adapt the webinar's content to address identified staff needs or implementation barriers we directly observe through visits and online diaries. This will engage staff in customizing the implementation support they receive. The webinars will be open to any interested clinic staff from Arms 2-3.

Arm 3 ('High' intensity support) components: All components as in Arm 2, plus PRACTICE FACILITATION site visits from the study team 'implementation specialist.' Visits will last 2-3 days, with 2 or more visits in implementation year 1, and 3 or more over the course of implementation years 2-3. The specialist will provide support as needed; anticipated activities include staff presentations, observational coaching on how the tools are presented to clinic staff and used in the clinic workflow, and tailored problem-solving support to help address identified barriers. Clinical questions arising at these visits will be fielded by our RN practice facilitator, and the site clinician champion. Advisory group clinicians will be asked to provide further support if needed.

#### 5. Study Population

#### a. Number of Subjects

Quantitative: 30 CHCs will be randomized to receive low, medium, or high-intensity support in implementing the ALL Initiative.

Qualitative: Study clinic providers and staff at OCHIN will participate in qualitative data collection efforts as described below.

#### b. Inclusion and Exclusion Criteria

Describe how individuals will be screened for eligibility and the criteria that define who will be included or excluded in your final study sample.

Describe the plan for disposition of data collected during recruitment/screening in the event of a screen failure or when a potential subject is contacted but declines participation (e.g. destroyed immediately, destroyed at end of study, retained for separate analysis or so that subjects are not contacted repeatedly about participation after they have declined, etc.)

#### Inclusion criteria.

Quantitative data: ~20,000 OCHIN patients from 30 clinics. Data will be extracted monthly from OCHIN's EHR including (a) Study population identification (age, CVD / DM, prescriptions); (b) Patient and (c) Clinic characteristics; (d) Patient outcomes (last BP, LDL results and measurement dates; issued prescriptions and dates); and (e) Process measures (e.g., tool use, encounters). (f) Cost analysis data will be collected as well.

<u>Qualitative data:</u> Ongoing phone calls with 30 point people. Site Visits: 18 visits in total. Breakdown: 6 clinics per year X 3 years. Interviews: 208 in total. We anticipate 108 formal (Breakdown: 6 clinics X 18 interviews) and 100 telephone (6 clinics X 12 interviews, plus 28 follow-up interviews).

Exclusion. Pregnant and lactating women will be excluded, as the ALL medications are contraindicated for pregnancy.

# c. Vulnerable Populations

**Regulatory Categories:** Indicate whether you will include or exclude each of the following populations. This refers to subjects who are known members of these populations upon recruitment or at any time during the study. You may not include members of these populations unless you describe this in your inclusion criteria.

- Children
- Pregnant women
- Neonates of uncertain viability or nonviable neonates (up to 28 days post birth)
- Prisoners (NOTE: The KPNW IRB does not have the appropriate membership to review research involving prisoners. Consultation with KFRI will be required.)

Justify the inclusion of any of these populations. Describe additional safeguards to protect the rights and welfare of these subjects.

Neonates (i.e., newborns) of uncertain viability or nonviable: Exclude

Children: Exclude

Decisionally/cognitively impaired: Include

Economically/educationally disadvantaged: Include

Non-English Speakers: Include

Employees who are specifically and intentionally targeted to be included in this study population because of

their workplace and/or employee status: Include

Elderly: Include

Prisoners: Prisoners are excluded or not anticipated to become study subjects

#### d. Setting

Describe the sites or locations where your research team will conduct the research.

*If this is a multi-site study:* 

- Specify what procedures are being performed at this site or by this site's personnel (consider recruitment, consent process, study procedures, data analysis, etc.).
- State how each site will satisfy its IRB review requirements. Indicate if you are asking this site's IRB to rely on another IRB or if another institution would like to rely on this site's IRB and include this information in the eIRB IRQ.

OCHIN member clinics (29 total): Winding Waters, Scappoose / OHSU, Santa Cruz County, Mosaic, Community HealthNet, Progressive Community Health Center, Truckee Tahoe Medical Group, Monterey Health Department, La Pine, Placer County, SW Montana, Neighborhood Family Practice

Michigan State University (MSU)

Mid-Atlantic Permanente Research Institute (MAPRI) – KPMAS

# e. Recruitment Methods

 Revised: 6.2.2016

Describe in detail how study participants will be recruited and enrolled. For example, will you openly recruit through the use of advertisements, websites, or brochures? Will you do targeted recruitment through the use of existing records or referral? If you will contact potential participants for recruitment, include the method(s) of contact and number of contact attempts that may be made.

Upload in the eIRB all recruitment materials, including brochures, advertisements, mailings, scripts, and website materials (screen shots). **Note:** If your materials are yet to be developed, these must be submitted to the IRB as a modification request and approved prior to use with study participants.

Describe, by position / title, who will be recruiting and enrolling participants (providing the particular names of research team members is not necessary).

Investigators sometimes plan to re-contact and re-recruit participants for future follow-up studies. That is, investigators may anticipate that participants for a currently proposed study will be logical participants in a future study. If there are any such expectations or plans for the participants in the currently proposed study to be re-contacted for follow-up studies, describe this. (And, note that participants should be informed of this potential for re-recruitment during the current study's consent process.)

Clinic recruitment will be led by Chris Nelson (Co-I) at OCHIN. Chris will follow-up with each clinic (who agreed to participate in the study during the proposal stage) by sending them an introductory email, FAQ handout and MOU. Patient data will be identified by the OCHIN DM registry. Staff and providers will be recruited by each OCHIN clinic's point person, specifically looking for local opinion leaders and / or as having strong positive or negative feelings about the intervention and support strategies used.

#### f. Consent Process

Describe how you will obtain and document consent, including:

- Where, when and how the consent process will take place.
- A process to ensure ongoing consent.
- Steps that will be taken to minimize the possibility of coercion or undue influence. Any steps that will be taken to ensure the subjects' understanding.

This research will use a consent procedure which does not include, or which alters, some or all of the elements of informed consent; or waives the requirement to obtain informed consent in its entirety. We are requesting a waiver of informed consent in its entirety for the quantitative and qualitative aspects of this study.

All of the following four statements are true: The research involves no more than minimal risk to the subjects; The waiver or alteration will not adversely affect the rights and welfare of the subjects; The research could not practicably be carried out without the waiver or alteration; and Whenever appropriate, the subjects will be provided with additional pertinent information after participation.

Explanation of Minimal Risk Research: Quantitative data (OCHIN patient data): OCHIN's EHR will be a Limited Data Set and will not include PHI. Data collection will not affect patients. Qualitative data (OCHIN providers and staff): Regular phone calls, site visits and interviews will include questions regarding views of the ALL initiative implementation, and not about individuals' health. Data collection will not affect providers or staff.

Explanation of Waiver or Alteration of Informed Consent: The waiver or alteration of informed consent will not adversely affect the rights and welfare of the subjects.

 Revised: 6.2.2016

Quantitative data (OCHIN patient data): consenting participants would require the release of full PHI rather than a LDS, therefore increasing their risk.

Qualitative data (OCHIN providers and staff): Obtaining consent would interfere with the clinic workflow

### **Modifications to the Consent Process**

- If you will not obtain consent or if you will be using only an abbreviated consent, explain how this will not
  adversely affect the rights and welfare of the subjects, why it is not practicable to obtain full consent,
  and, if appropriate, what additional pertinent information will be provided to subjects after
  participation.
  - <u>Example 1</u>: If part of your study involves retrospective review of existing data for many individuals, it may not be practicable to collect the data you need if you had to contact each individual to get permission. As long as confidentiality of the information is protected, such data collection poses minimal risk to the subjects and would not adversely impact their rights or welfare.)
  - <u>Example 2:</u> Studies that require 100% participation in order to obtain valid results, such as studies where an entire clinic is randomized to participate in an intervention, may not be practicable to conduct if informed consent is required.
- If you will conduct screening or any other research procedures before obtaining full informed consent, describe this and explain how the above criteria are met with respect to that part of the study.

# **Non-English Speaking Subjects**

- If subjects who do not speak English will be enrolled, describe how the consent discussion will take place and indicate if translated consent forms or short forms will be used.
- Confirm that an interpreter will assist with the initial consent process and subsequent study visits.

#### Assent of Children and Parent Permission

- Describe your plan for obtaining parent permission. The permission of one parent is generally sufficient for minimal risk research, or for greater than minimal risk research if there is the potential for direct benefit to the child.
- Note that for studies involving greater than minimal risk with no prospect of direct benefit to the child subjects, permission of both parents is required unless one parent is deceased, unknown, incompetent, or not reasonably available, or when only one parent has legal responsibility for the care and custody of the child.
- Describe whether permission will be obtained from individuals other than parents, and if so, who will be allowed to provide permission.
- Indicate whether assent will be obtained and documented from all, some, or none of the children. If assent will only be obtained from some children (because of very young age, severe cognitive impairment, etc.), indicate which children will be required to assent and which will not.
- When assent of children is obtained, describe whether and how it will be documented.
- When subjects might reach the age of majority during the study, describe the plan to obtain consent from these subjects at that time using an adult consent form.

# Adults Unable to Consent/Decisionally Impaired

Describe the process to determine whether an individual is capable of consent.

 Revised: 6.2.2016

- List the individuals from whom permission will be obtained in order of priority. (E.g., durable power of attorney for health care, court appointed guardian for health care decisions, spouse, and adult child. See the KPNW Policy on Surrogate Consent for Research for more information.)
- Describe the process for assent of the subjects. Address the following:
  - Whether assent will be required of all, some, or none of the subjects. If assent will be obtained from some subjects, indicate which subjects will be required to assent and which will not.
  - If assent will not be obtained from some or all subjects, an explanation of why not.
  - o When assent is obtained, describe how it will be documented.
- Describe the plan to obtain consent if subjects might regain capacity to consent during the study.

# HIPAA Privacy Rule Authorization – if study will use or disclose Protected Health Information (PHI)

- Describe the plan to obtain a signed Privacy Rule Authorization from each subject.
- If you will not obtain signed Privacy Rule Authorization or if you want to eliminate any required language from the authorization, explain:
  - Why the research could not practicably be conducted without the waiver or alteration (for example, you may not be able to do the research, or part of the research, if you needed to contact each individual for permission because of lack of contact information or a large number of individuals);
  - Why access to and use of the PHI is necessary for the research; and
  - O Why the use or disclosure of PHI for the research poses no greater than minimal risk to the subjects' privacy (must have an adequate plan to protect the PHI from improper use or disclosure, a plan to destroy identifiers at the earliest opportunity consistent with the purpose of the research, and, when applicable, written assurances from collaborators that PHI will not be reused or re-disclosed to any other entity).

Not applicable.

# 6. Study Procedures

Describe:

- All research procedures being performed and when they are performed, including timing and amount of all samples collected for research purposes.
- Measures taken to lessen the probability or magnitude of risks (monitoring for safety, preventing complications, etc.).
- All drugs and devices used in the research and the purpose of their use, and their FDA approval status.
- Data collection tools (upload all surveys, scripts, and data collection forms).
- What data will be collected, including long-term follow-up.
- The duration of an individual subject's participation in the study.

**NOTE:** It should be clear exactly which procedures will be conducted for the research as opposed to procedures the subjects would undergo (in the exact manner described in the protocol) even if they were not participating in the study.

Describe procedures that will be followed when subjects withdraw from the research, including withdrawal from intervention but continued data collection.

Describe any anticipated circumstances under which subjects will be withdrawn from the research without their consent.


If the study involves genetic testing or collection of genetic information, describe this.

If the study involves **anonymous or coded genetic research and consent for genetic research will NOT be obtained**, confirm here that you will check the genetic exclusions database in order to comply with the Oregon Genetic Privacy Law.

#### Qualitative data:

**The All Staff Survey.** All staff at the SPREAD-NET (S-N) study clinics (~30 anticipated) will be asked to complete this paper survey, which is designed to assess each clinic's readiness to change.

**Clinic Information Form (CIF) Survey.** One person, e.g., clinic manager or quality improvement coordinator, at each of the study clinics will be asked to complete a paper survey which is intended to collect factual information about the clinic that will be used to help understand how best to support implementation of the ALL Initiative.

**Bi-weekly phone calls with point people.** Once the ALL initiative has been implemented in the study clinics (estimated March 2015), each clinic's study point person will participate in regular telephone calls with study staff at KPCHR and OCHIN. These calls will be biweekly to start; the number of calls per month may taper off over time. Calls are expected to last 15- 30 minutes. No PHI will be collected, nor will data be collected from or about patients. The format of the calls will be fairly unstructured; in general study staff will solicit information on barriers and facilitators to the uptake of the ALL initiative, including use of the study tools and fit into clinic workflows. The attached 'Topics for point person calls' document lists subjects that may be covered during these calls. Phone calls will be recorded by study staff using KPCHR-approved digital recorders that are encrypted and password protected for security and confidentiality, and transcribed by a KPCHR approved transcriptionist as necessary. Recordings and transcripts will be sent through KPCHR's secure file transfer site.

**Site visits.** In study years 2.5-4, we will conduct in-person observations at 6 clinics per year, to collect in-depth data to augment the data collected in the diary entries. We will purposively select CHCs for site visits that will optimize our learning, such as CHCs that are excelling with lower levels of support. At each visit, 2 members of our qualitative team will spend 2 days at the CHC. Ethnographic methods (field observation, opportunistic and semi-structured interviews) will be used. Such methods are uniquely suited to the study of organizational behavior as they facilitate indepth understanding of change processes, workflows and routines, and barriers and facilitators to change. At these visits, we will explore the implementation process, toolkit use and barriers and enablers of practice change, including understanding clinic workflow for DM / CVD patients, and how ALL supports medication decision-making.

**Additional interviews.** In years 3-4.5, our qualitative team will conduct telephone or video-based semi-structured interviews with staff at each CHC that we do not visit in person. The interviews will be designed to elicit further information about how ALL was implemented, how effectively each arm's strategy supported that implementation, and barriers to effectiveness. We will also likely conduct more informal, follow-up interviews to fill in knowledge gaps identified during subsequent data collection and analysis.

Other qualitative data sources. Our team will also collect 'archival' data related to the process evaluation (e.g., email / telephone discussions with CHC staff; clinic policies; concurrent QI initiatives, as well as conduct regular debriefings with practice facilitators (arm 3)).

Quantitative data: This data will be extracted monthly from OCHIN's EHR will include: (a) Study population identification (age, CVD / DM, prescriptions); (b) Patient and (c) Clinic characteristics; (d) Patient outcomes

 Revised: 6.2.2016

(last BP, LDL results and measurement dates; issued prescriptions and dates); and (e) Process measures (e.g., tool use, encounters). Cost data will be collected as well.

# 7. Data Analysis

# a. Analysis Plan

Describe the data analysis plan, including any statistical procedures.

When applicable, provide a power analysis.

Describe any procedures that will be used for quality control of collected data.

Survey data analyses. Survey results will be used for two purposes. (1) Summary results will be used as a 'diagnostic tool' to identify materials needed to train Arm 2-3 clinics at the in-person training and subsequent webinars. We will use descriptive statistics to summarize the responses to the surveys and identify prevalent aspects to be included in the trainings. (2) Results will be used to measure the clinics' baseline characteristics, which will be included in longitudinal analyses as covariates. We will test for baseline differences in patient and clinic characteristics between study arm clinics using chi-square and t-tests to determine if differences exist. Qualitative survey results from open-ended questions will be content-analyzed by our qualitative team using standard methods<sup>225,226</sup>

Specific Aim 1 & 2 analyses. For Aim 1, we will use an interrupted time-series design with threelevel hierarchical linear models to assess differences in the impact of the intervention's implementation, across the 3 support strategies, on quantitative outcomes (patient health [Effectiveness], guideline-based prescribing [Reach]). This method is commonly used to compare changes in rates across time pre- and post- implementation. Time in monthly intervals will form the 1st level of the model, person the 2nd, and clinic the 3rd; these models do not require patient-level data at all time points. We will include a dummy-coded variable for study arm (reference group = 'High'-intensity support) and clinic level covariates (as guided by the Practice Change Model components) at model level-3, and patient level covariates at level-2. The level-1 model will be specified as a segmented regression model, to yield an estimate of the level and slope across time of rate of the outcomes of interest in the 2 years pre-implementation, and changes in the level and slope of these rates in the 12 months post-implementation. Change in level provides an estimate of the immediate effect of the intervention. Change in slope gives an estimate of effect across time. We will include a cross-level interaction of study arm with time, change in level, and change in slope; the interaction of change in slope by study arm tests if the change from pre to post intervention in the trends in the rates over time differs across arms. Similarly, the interaction of change in level by study arm tests if the immediate effect of the intervention differs across study arms. Separate analyses will be conducted for percent of patients with guideline-appropriate prescriptions for ACE/ARBs, statins (our primary outcomes), and with last BP under control, and last LDL under control (secondary outcomes) (Table 5). Aim 2 analyses will use the same approach, adding time points through 36 months post-intervention [Maintenance]. The time period variable will have 3 levels (pre-intervention, 12 months post-, and 13-36 months post-intervention). Of interest is whether the slopes (rate of change) or level in the last time period differ across the 3 arms.

Statistical power. Segmented regression is a powerful statistical technique in diverse applications, but formal power analyses may not be feasible as estimates of the model parameters are not available prior to the study. We will meet or exceed the 12 points pre- and post-intervention used in similar segmented regression analyses, as is adequate to detect even modest effect. To illustrate our power to detect changes between study arms, we conducted a


power analysis using data from our current study. At 12 months post-intervention, 60%, 63% and 46% of control clinic patients and 68%, 76%, and 58% of intervention clinic patients were appropriately on statins, ACE, and both, respectively. We can detect differences of this magnitude between any two arms of the study with power of .95 to .99 if the intra-class correlation is .01, and power of .76 to .99 if the ICC is .02 with an alpha level of .05.

Additional analyses (Minimal support needed to achieve treatment thresholds): While our primary analyses will measure implementation impact as described above, we will also conduct secondary analyses, for both the patient health and guideline-based prescribing outcomes, in which we will define thresholds of intervention impact. Thresholds will be defined as a target percentage of clinic patients with (i) guideline-appropriate prescriptions; (ii) last LDL <100; and (iii) last systolic BP <135. Targets will be determined based on baseline data and in consultation with the SPREAD-NET advisory group, which includes CHC clinicians. We will then assess the minimal amount of implementation support needed to achieve threshold results. We anticipate based on our first study that these targets will be approximately (i) 75%; (ii) 70%; and (iii) 80%, respectively. Logistic regression will be used, with study arm (reference group = High support) predicting a binary outcome for threshold achieved by 12 months.

Qualitative analyses (Aim 3). Led by Dr. Cohen, our expert qualitative team will analyze data from the weekly diaries, site visits, archival data, observation, and interviews, to gain in-depth knowledge of the change process. Data collection and analyses will be concurrent and iterative, permitting us to identify salient constructs and knowledge gaps while implementation is ongoing, incorporate this knowledge into subsequent data collection, and guide adaptation of the support strategies. A grounded theory approach coupled with an immersion-crystallization process will be used to identify themes and patterns in the qualitative data. The aim will be to understand what happens during implementation from the participants' perspective, including barriers and facilitators, the extent to which toolkit elements are used or adapted [Adoption], and the impact of each support strategy on implementation success [Implementation]. Particular attention will be paid to factors leading to a given practice excelling or struggling in response to the offered implementation support. Our team will use Miller and Crabtree's 5-phase analysis strategy, as team members have previously done successfully.

# b. Sharing of Results with Subjects

Describe whether results (study results or individual subject results, such as results of standard or research lab tests and genetic tests) will be shared with subjects or their providers.

If the study carries a risk of incidental findings, describe your plan for evaluating these and determining whether and how subjects or their providers will be given this information.

If laboratory results will be shared with subjects or their healthcare providers, verify that the laboratory conducting the test is CLIA certified.

Not applicable.

#### c. Data and Specimen Banking

Indicate if specimens may be used for future research and whether that may include genetic research (see above regarding requirements for anonymous or coded genetic research).

State if data or specimens will be sent to a separate repository.


Revised: 6.2.2016

If data or specimens will be banked in a repository for future use as part of this protocol submission, describe here (or in a separate document) where they will be stored, how long they will be stored, how they may be accessed, and who will have access to the specimens. Describe the procedures to release data or specimens, including: the process to request a release, approvals required for release, who can obtain data or specimens, and the data to be provided with specimens.

Not applicable.

# 8. Privacy, Confidentiality, and Data Security

Describe the steps that will be taken to protect subjects' privacy during recruitment, consent and study procedures.

Describe the plan for storage of data and specimens, including:

- Where the materials will be stored.
- How the materials will be labeled.
- Any other steps that will be taken to ensure security (e.g., training of staff, authorization of
  access, password protection, encryption, physical security, and separation of identifiers from
  data and specimens, certificates of confidentiality).
- Plan to destroy/archive or retain data and/or specimens at the end of the study.

If you will collect any data from participants electronically (including email, website, etc.), explain:

- How the data will be collected.
- How the information will be secured (encryption, password protection, etc.; may require consultation with IT department).
- Any risks to the participants' privacy posed by using these methods (describe in consent, as applicable).
- How you will verify the participant's identity.

If any data or specimens will be sent outside of this site, list each recipient (may list by role or category if the information is the same for several different entities). For each recipient, describe:

- What will be sent.
- Whether the materials will be fully identifiable (PHI, if health information), a Limited Data Set, de-identified, or aggregate (See <u>Types of Compliance Data – Quick Reference</u> for more information).
- How the materials will be transferred securely (for instance, Secure File Transfer).
- NOTE: If you are sending full PHI outside this site, you must have a RAMP review. Complete and upload the <u>Risk Assessment Tool</u>.

Quantitative data: This will be stored at OCHIN. Qualitative data: This will be stored at CHR.

CHR investigators and project staff sign annual confidentiality pledges and receive IRB training and Certification every three years. Data from the community clinics will come through OCHIN, and OCHIN will use similar safeguards to ensure confidentiality when handling data. OCHIN will use unique patient identification codes and all data sources will be linked through a secure relational database at OCHIN. Data will only be shared with CHR through a secure data transfer web site. After data have been linked and transferred, they will be de-identified for analytical purposes. OCHIN and CHR will use a state-of-the art file transfer application to provide secure file transfers. This application transfers data from a secured sending website to a secured receiving website. CHR's standards meet the standards required f


or DHHS level 1 security. In addition, back-end checks will be conducted periodically to *ensure data* reliability.

# 9. Provisions to Monitor the Data to Ensure the Safety of Subjects

This is required when research involves more than Minimal Risk to subjects. Describe:

- Who will monitor the study data for safety.
- Who will verify data accuracy and conduct quality assessments.
- How objectivity in the monitoring process will be ensured.
- What data and/or events will be reported to the monitor or monitoring board and how frequently.
- The procedures and methods that the monitor or board will use to evaluate the data.
- Criteria for taking action on monitoring findings (for instance, stopping rules, reporting, protocol changes, changes to monitoring frequency or plan).
- For studies monitored by a DSMB/C, describe the committee membership and structure, meeting format, and quorum requirements. Upload the board/committee charter, if one exists.

# 10. Risks and Benefits

#### a. Risks to Subjects

List the reasonably foreseeable risks, discomforts, hazards, or inconveniences to the subjects related the subjects' participation in the research. Describe the probability, magnitude, duration, and reversibility of the risks. Consider physical, psychological, social, legal, and economic risks.

Risk of breach of confidentiality is common to almost all research studies. Avoid indicating that study participation is expected to be "risk-free" or without risk.

If applicable, indicate which procedures may have risks to the subjects that are currently unforeseeable.

If applicable, indicate which procedures may have risks to an embryo or fetus should the subject be or become pregnant.

If applicable, describe risks to others who are not subjects and risks to Kaiser Permanente.

### b. Potential Benefits to Subjects

Describe the potential benefits that individual subjects may experience from taking part in the research. Include the probability, magnitude, and duration of the potential benefits.

Indicate if there is no direct benefit. Do not include benefits to society or others.

**Note:** Compensation is not considered a benefit and should not be included in this section. See Compensation to Participants section.

### 11. Costs to Participants

Describe any costs that participant may be responsible for due to participating in this study (for example, co-pays; paying for treatment, therapies, or other interventions, or the delivery of these) and how you will inform participants of these costs prior to their enrollment in this study.

 Revised: 6.2.2016

# 12. Compensation to Participants

Describe any compensation provided to participants, for example, for time inconvenience, discomfort, travel, or in the event of research related injury.

If applicable, describe how you will inform participants of this prior to their enrollment in the study, including if payment will be prorated if the subject withdraws early from the study.

**Note:** payment may not be withheld as an incentive for participants to complete the study.

# 13. Resources Available (delete if not applicable)

Describe any special resources or expertise required to conduct the study.

# 14. Drugs or Devices (delete if not applicable)

If the research involves drugs or devices and is investigator-initiated, indicate whether there is any possibility that the results will be reported to FDA (e.g. as part of a new drug application [NDA] or premarket approval application [PMA]).

If this is a device study and you think the device is Non-Significant Risk, include justification here or upload it as a separate document along with any available device information (instructions for use, etc.).

If the drug is investigational (has an IND) or the device has an IDE or a claim of abbreviated IDE (Non-Significant Risk device), confirm that you will comply with all applicable FDA requirements for investigators. Also see the <u>ICH-GCP guidance</u> for a summary of investigator and sponsor responsibilities in clinical trials.

Address the items listed below as applicable.

#### **Drug Studies:**

- Confirm that you will follow applicable KP pharmacy policies and procedures.
- Describe your plan for drug storage, handling, and accountability, including distribution, return, and destruction of the drug(s).
- If applicable, upload a copy of the Investigator Brochure for each drug. (If this is not an Oncology study, you must also send an additional copy to the Regional Formulary and Therapeutics Committee.)

#### Device Studies:

- Describe the device, the manufacturing process, and the device labeling, including safety instructions or warnings. If available, this may be addressed in separately uploaded device information (such as instructions for use).
- Describe device storage, handling, and accountability, including how access to the device will be limited to appropriate personnel and how you will ensure the device will be used only for appropriate study subjects.

# 15. Multi-Site Coordination (delete if not applicable)

If this site will be the coordinating center for any activities, describe those activities here or in a separate document.

Describe the processes to ensure communication among sites, such as:

- All sites have the most current version of the protocol, consent document, and HIPAA authorization.
- All required approvals have been obtained at each site (including approval by the site's IRB of record).
- All modifications have been communicated to sites, and approved (including approval by the site's IRB of record) before the modification is implemented.
- All engaged participating sites will safeguard data as required by local information security policies.
- All local site investigators conduct the study appropriately.
- All non-compliance with the study protocol or applicable requirements will reported in accordance with local policy.
- Communication of problems, interim results, and study closure.

# 16. Community-Based Participatory Research (delete if not applicable)

Describe involvement of the community in the design and conduct of the research.

Describe your plan for ensuring that community research partners are appropriately trained in human subjects protection.

**NOTE:** "Community-based Participatory Research" is a collaborative approach to research that equitably involves all partners in the research process and recognizes the unique strengths that each brings. Community-based Participatory Research begins with a research topic of importance to the community, has the aim of combining knowledge with action and achieving social change to improve health outcomes and eliminate health disparities.


# Bibliography and References Cited

- 1. Mendel P, Meredith LS, Schoenbaum M, Sherbourne CD, Wells KB. Interventions in organizational and community context: a framework for building evidence on dissemination and implementation in health services research. *Adm Policy Ment Health* 2008 Mar; 35(1-2):21-37.
- 2. Glasgow RE, Emmons KM. How can we increase translation of research into practice? Types of evidence needed. *Annu Rev Public Health* 2007; 28:413-33.:413-433.
- 3. Rubenstein LV, Pugh J. Strategies for promoting organizational and practice change by advancing implementation research. *J Gen Intern Med* 2006 Feb; 21 Suppl 2:S58-64.:S58-S64.
- 4. Godley SH, Garner BR, Smith JE, Meyers RJ, Godley MD. A large-scale dissemination and implementation model for evidence-based treatment and continuing care. *Clin Psychol (New York)* 2011 Mar; 18(1):67-83.
- 5. Greenhalgh T, Robert G, Macfarlane F, Bate P, Kyriakidou O. Diffusion of innovations in service organizations: systematic review and recommendations. *Milbank Q* 2004; 82(4):581-629.
- 6. Lanham HJ, Leykum LK, Taylor BS, McCannon CJ, Lindberg C, Lester RT. How complexity science can inform scale-up and spread in health care: Understanding the role of self-organization in variation across local contexts. Soc Sci Med 2012 Jul 4. [Epub ahead of print]
- 7. Katz DL, Murimi M, Gonzalez A, Njike V, Green LW. From controlled trial to community adoption: the multisite translational community trial. *Am J Public Health* 2011 Aug; 101(8):e17-e27.
- 8. Harris JR, Cheadle A, Hannon PA, Forehand M, Lichiello P, Mahoney E, Snyder S, Yarrow J. A framework for disseminating evidence-based health promotion practices. *Prev Chronic Dis* 2012; 9:E22. Epub@2011 Dec 15.:E22.
- 9. Wandersman A, Duffy J, Flaspohler P, Noonan R, Lubell K, Stillman L, Blachman M, Dunville R, Saul J. Bridging the gap between prevention research and practice: the interactive systems framework for dissemination and implementation. *Am J Community Psychol* 2008 Jun; 41(3-4):171-181.
- 10. Glasgow RE, Vinson C, Chambers D, Khoury MJ, Kaplan RM, Hunter C. National Institutes of Health approaches to dissemination and implementation science: current and future directions. *Am J Public Health* 2012 Jul; 102(7):1274-1281.
- 11. Simmons R, Fajans P, Ghiron L. Scaling up health service delivery: from pilot innovations to policies and programmes. Geneva: The World Health Organization. Available at: https://extranet.who.int/iris/restricted/bitstream/10665/43794/1/9789241563512\_eng.pdf. Accessed on: 1-9-2013.
- 12. Nieva VF, Swift E, Fair S. AHRQ Health Care Innovations Exchange report on Scale up and Spread Activities 2011. AHRQ Report, 2011. 2011.
- 13. Dingfelder HE, Mandell DS. Bridging the research-to-practice gap in autism intervention: an application of diffusion of innovation theory. *J Autism Dev Disord* 2011 May; 41(5):597-609.
- Cilenti D, Brownson RC, Umble K, Erwin PC, Summers R. Information-seeking behaviors and other factors contributing to successful implementation of evidence-based practices in local health departments. J Public Health Manag Pract 2012 Nov; 18(6):571-576.
- 15. Powell BJ, McMillen JC, Proctor EK, Carpenter CR, Griffey RT, Bunger AC, Glass JE, York JL. A compilation of strategies for implementing clinical innovations in health and mental health. *Med Care Res Rev* 2012 Apr; 69(2):123-157.
- 16. US Department of Health & Human Services. U.S. Department of Health & Human Services Strategic Plan Fiscal Years 2010 2015. Available at: <a href="http://www.hhs.gov/secretary/about/priorities/strategicplan2010-2015.pdf">http://www.hhs.gov/secretary/about/priorities/strategicplan2010-2015.pdf</a>. Accessed on: 1-24-2013.
- 17. Dudl RJ, Wang MC, Wong M, Bellows J. Preventing myocardial infarction and stroke with a simplified bundle of cardioprotective medications. *Am J Manag Care* 2009 Oct 1; 15(10):e88-e94.
- 18. Gold R, Muench J, Turner A, Mital M, Milano C, Shah A, Nelson C, DeVoe JE, Nichols G. Collaborative development of a randomized study to adapt a diabetes quality improvement initiative for federally

- qualified health centers . *Journal of Health Care for the Poor and Underserved* 2012 Aug; 23(3 Suppl):236-246.
- 19. Gold R, Nichols G, Muench J, Hill C, Mital M, Dudl J, DeVoe J, Puro J, Nelson C. Implementing an Integrated Care Setting's Diabetes QI Initiative in Safety Net Clinics: A Practice-Based Randomized Trial. Oral presentation: March 2012 at the 5<sup>th</sup> Annual NIH conference on the Science of Dissemination and implementation: Science at the Crossroads. Bethesda, MD. 2012 Mar 20.
- 20. Gold R, Meunch J, Hill.C., Milano C, Turner A, Nelson C, Mital M, DeVoe J, Puro J. Can a Privately Developed Quality Improvement Initiative be Adapted for Implementation in Primary Care Safety Net Clinics? Oral presentation: December 2012 at the 40th Annual North American Primary Care Research Group conference. New Orleans, LA. 2012 Dec 5.
- 21. Durlak JA, DuPre EP. Implementation matters: a review of research on the influence of implementation on program outcomes and the factors affecting implementation. *Am J Community Psychol* 2008 Jun; 41(3-4):327-350.
- 22. Rohrbach LA, Gunning M, Sun P, Sussman S. The Project Towards No Drug Abuse (TND) dissemination trial: implementation fidelity and immediate outcomes. *Prev Sci* 2010 Mar; 11(1):77-88.
- 23. Woolf SH, Johnson RE. Erratum in The Project Towards No Drug Abuse (TND) dissemination trial: implementation fidelity and immediate outcomes. *Prev Sci* 2010 Mar; 11(1):113.
- 24. van de Steeg-van Gompel CH, Wensing M, De Smet PA. Implementation of adherence support for patients with hypertension despite antihypertensive therapy in general practice: a cluster randomized trial. *Am J Hypertens* 2010 Sep; 23(9):1038-1045.
- 25. Feldstein AC, Glasgow RE. A practical, robust implementation and sustainability model (PRISM) for integrating research findings into practice. *Jt Comm J Qual Patient Saf* 2008 Apr; 34(4):228-243.
- 26. Gaglio B, Glasgow R. Evaluation approaches for dissemination and implementation research. In: Brownson RCCGA, Proctor EK, eds. *Dissemination and Implementation Research in Health*. New York: Oxford, 2012.
- 27. Glasgow RE, Marcus AC, Bull SS, Wilson KM. Disseminating effective cancer screening interventions. *Cancer* 2004 Sep 1; 101(5 Suppl):1239-1250.
- 28. Glasgow RE, Goldstein MG, Ockene JK, Pronk NP. Translating what we have learned into practice. Principles and hypotheses for interventions addressing multiple behaviors in primary care. *Am J Prev Med* 2004 Aug; 27(2 Suppl):88-101.
- 29. Cohen D, McDaniel RR, Jr., Crabtree BF, Ruhe MC, Weyer SM, Tallia A, Miller WL, Goodwin MA, Nutting P, Solberg LI, Zyzanski SJ, Jaen CR, Gilchrist V, Stange KC. A practice change model for quality improvement in primary care practice. *J Healthc Manag* 2004 May; 49(3):155-168; discussion 169-170.
- 30. Kessler RS, Purcell EP, Glasgow RE, Klesges LM, Benkeser RM, Peek CJ. What Does It Mean to "Employ" the RE-AIM Model? *Eval Health Prof* 2012 May 21. [Epub ahead of print]
- 31. American Diabetes Association. Economic costs of diabetes in the U.S. in 2007. *Diabetes Care* 2008; 31(3):596-615.
- 32. Centers for Disease Control and Prevention. National Diabetes fact sheet: national estimates and general information on diabetes and prediabetes in the United States, 2011. Atlanta, GA:U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, 2011. Available at: <a href="http://www.cdc.gov/diabetes/pubs/pdf/ndfs">http://www.cdc.gov/diabetes/pubs/pdf/ndfs</a> 2011.pdf. Accessed on: 4-11-2012.
- 33. Mokdad AH, Ford ES, Bowman BA, Nelson DE, Engelgau MM, Vinicor F, Marks JS. The continuing increase of diabetes in the US. *Diabetes Care* 2001 Feb; 24(2):412.
- 34. Narayan KMV, Zhang P, Kanaya A, Williams D, Engelgau M, Imperatore G, Ramachandran A. Diabetes: the pandemic and potential solutions. In: Jamison JT, Breman JG, Measham AR, Alleyne G, Claeson M, Evans DB, Prabhat J, Mills A, Musgrove P, eds. *Disease Control Priorities in Developing Countries*. Washington DC: Oxford University Press, World Bank, 2006, pp 591-604.
- 35. Narayan KMV, Boyle JP, Geiss LS, Saaddine JB, Thompson TJ. Impact of recent increase in incidence on future diabetes burden: U.S., 2005-2050. *Diabetes Care* 2006 Sep; 29(9):2114-2116.

- 36. Boyle JP, Honeycutt AA, Narayan KM, Hoerger TJ, Geiss LS, Chen H, Thompson TJ. Projection of diabetes burden through 2050: impact of changing demography and disease prevalence in the U.S. *Diabetes Care* 2001 Nov; 24(11):1936-1940.
- 37. Nauta ST, Deckers JW, Akkerhuis KM, van Domburg RT. Short- and long-term mortality after myocardial infarction in patients with and without diabetes: changes from 1985 to 2008. *Diabetes Care* 2012 Oct; 35(10):2043-2047.
- 38. Mensah GA, Brown DW. An overview of cardiovascular disease burden in the United States. *Health Affairs* 2007; 26(1):38-48.
- 39. Nichols GA, Brown JB. The impact of cardiovascular disease on medical care costs in subjects with and without type 2 diabetes. *Diabetes Care* 2002 Mar; 25(3):482-486.
- 40. Davidson MH. Cardiovascular risk factors in a patient with diabetes mellitus and coronary artery disease: therapeutic approaches to improve outcomes: perspectives of a preventive cardiologist. *Am J Cardiol* 2012 Nov 6; 110(9 Suppl):43B-49B.
- 41. Egede LE, Gebregziabher M, Dismuke CE, Lynch CP, Axon RN, Zhao Y, Mauldin PD. Medication nonadherence in diabetes: Longitudinal effects on costs and potential cost savings from improvement. *Diabetes Care* 2012 Dec; 35(12):2533-2539.
- 42. Green LW, Ottoson JM, Garcia C, Hiatt RA. Diffusion theory and knowledge dissemination, utilization, and integration in public health. *Annu Rev Public Health* 2009; 30:151-74. doi: 10.1146/annurev.publhealth.031308.100049.:151-174.
- 43. Flaspohler P, Lesesne CA, Puddy RW, Smith E, Wandersman A. Advances in Bridging Research and Practice: Introduction to the Second Special Issue on the Interactive System Framework for Dissemination and Implementation. *Am J Community Psychol* 2012 Aug 9.
- 44. Tabak RG, Khoong EC, Chambers DA, Brownson RC. Bridging research and practice: models for dissemination and implementation research. *Am J Prev Med* 2012 Sep; 43(3):337-350.
- 45. Brownson RC, Colditz GA, Proctor EK (Eds). *Dissemination and Implementation Research in Health*. NY, NY: Oxford U Press; 2012.
- 46. American Diabetes Association. Standards of medical care in diabetes--2012. *Diabetes Care* 2012 Jan; 35 Suppl 1:S11-S63.
- 47. Antithrombotic Trialists' Collaboration. Collaborative meta-analysis of randomised trials of antiplatelet therapy for prevention of death, myocardial infarction, and stroke in high risk patients. *BMJ* 2002 Jan 12; 324(7329):71-86.
- 48. Baigent C, Keech A, Kearney PM, Blackwell L, Buck G, Pollicino C, Kirby A, Sourjina T, Peto R, Collins R, Simes R. Efficacy and safety of cholesterol-lowering treatment: prospective meta-analysis of data from 90,056 participants in 14 randomised trials of statins. *Lancet* 2005 Oct 8; 366(9493):1267-1278.
- 49. Brenner BM, Cooper ME, de Zeeuw D, Keane WF, Mitch WE, Parving HH, Remuzzi G, Snapinn SM, Zhang Z, Shahinfar S. Effects of losartan on renal and cardiovascular outcomes in patients with type 2 diabetes and nephropathy. *N Engl J Med* 2001 Sep; 345(12):861-869.
- 50. Cholesterol Treatment Trialists (CCT) Collaborators. Efficacy of cholesterol-lowering therapy in 18,686 people with diabetes in 14 randomised trials of statins: a meta-analysis. *Lancet* 2008; 371:117-125.
- 51. Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. *Lancet* 2010 Nov 13; 376(9753):1670-1681.
- 52. Collins R, Armitage J, Parish S, Sleigh P, Peto R. MRC/BHF Heart Protection Study of cholesterol-lowering with simvastatin in 5963 people with diabetes: a randomised placebo-controlled trial. *Lancet* 2003 Jun 14: 361(9374):2005-2016.
- 53. Daly CA, Fox KM, Remme WJ, Bertrand ME, Ferrari R, Simoons ML. The effect of perindopril on cardiovascular morbidity and mortality in patients with diabetes in the EUROPA study: results from the PERSUADE substudy. *Eur Heart J* 2005 Jul; 26(14):1369-1378.
- Downs JR, Clearfield M, Weis S, Whitney E, Shapiro DR, Beere PA, Langendorfer A, Stein EA, Kruyer W, Gotto AM, Jr. Primary prevention of acute coronary events with lovastatin in men and women with

- average cholesterol levels: results of AFCAPS/TexCAPS. Air Force/Texas Coronary Atherosclerosis Prevention Study. *JAMA* 1998 May 27; 279(20):1615-1622.
- 55. Fox KM. Efficacy of perindopril in reduction of cardiovascular events among patients with stable coronary artery disease: randomised, double-blind, placebo-controlled, multicentre trial (the EUROPA study). *Lancet* 2003 Sep 6; 362(9386):782-788.
- 56. Fox KM, Bertrand ME, Remme WJ, Ferrari R, Simoons ML, Deckers JW. Efficacy of perindopril in reducing risk of cardiac events in patients with revascularized coronary artery disease. *Am Heart J* 2007 Apr; 153(4):629-635.
- 57. Gaede P, Vedel P, Larsen N, Jensen GV, Parving HH, Pedersen O. Multifactorial intervention and cardiovascular disease in patients with type 2 diabetes. *N Engl J Med* 2003 Jan 30; 348(5):383-393.
- 58. Hayward RA, Hofer TP, Vijan S. Narrative review: Lack of evidence for recommended low-density lipoprotein treatment targets: A solvable problem. *Ann Intern Med* 2006 Oct; 145:520-530.
- 59. HOPE. Effects of ramipril on cardiovascular and microvascular outcomes in people with diabetes mellitus: results of the HOPE study and MICRO-HOPE substudy. Heart Outcomes Prevention Evaluation Study Investigators [see comments]. *Lancet* 2000 Jan 22; 355(9200):253-259.
- 60. Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol lowering with simvastatin in 20,536 high-risk individuals: a randomised placebo-controlled trial. *Lancet* 2002 Jul 6; 360(9326):7-22.
- 61. Farmer JA, Gotto AM, Jr. The Heart Protection Study: expanding the boundaries for high-risk coronary disease prevention. *Am J Cardiol* 2003 Jul 3; 92(1A):3i-9i.
- 62. Klausen K, Borch-Johnsen K, Jensen G, Clausen P, Scharling H, Appleyard M, Jensen JS. Very low levels of microalbuminuria are associated with increased risk of coronary heart disease an death independent of renal function, hypertension, and diabetes. *Circulation* 2004; 110:32-35.
- 63. Law MR, Wald NJ, Rudnicka AR. Quantifying effect of statins on low density lipoprotein cholesterol, ischaemic heart disease, and stroke: systematic review and meta-analysis. *BMJ* 2003 Jun 28; 326(7404):1423.
- 64. LIPID Study Group. Prevention of cardiovascular events and death with pravastatin in patients with coronary heart disease and a broad range of initial cholesterol levels. *New England Journal of Medicine* 1998; 339(19):1349-1357.
- 65. Heart Protection Study Collaborative Group. MRC/BHF Heart Protection Study of cholesterol-lowering therapy and of antioxidant vitamin supplementation in a wide range of patients at increased risk of coronary heart disease death: early safety and efficacy experience. *Eur Heart J* 1999 May; 20(10):725-741.
- 66. Pedersen TR, Wilhelmsen L, Faergeman O, Strandberg TE, Thorgeirsson G, Troedsson L, Kristianson J, Berg K, Cook TJ, Haghfelt T, Kjekshus J, Miettinen T, Olsson AG, Pyorala K, Wedel H. Follow-up study of patients randomized in the Scandinavian simvastatin survival study (4S) of cholesterol lowering. *Am J Cardiol* 2000 Aug 1; 86(3):257-262.
- 67. PROGRESS Collaborative Group. Randomised trial of a perindopril-based blood-pressure-lowering regimen among 6,105 individuals with previous stroke or transient ischaemic attack. *Lancet* 2001 Sep 29; 358(9287):1033-1041.
- 68. Pyorala K, Pedersen TR, Kjekshus J, Faergeman O, Olsson AG, Thorgeirsson G. Cholesterol lowering with simvastatin improves prognosis of diabetic patients with coronary heart disease. A subgroup analysis of the Scandinavian Simvastatin Survival Study (4S) [see comments] [published erratum appears in Diabetes Care 1997 Jun;20(6):1048]. *Diabetes Care* 1997 Apr; 20(4):614-620.
- 69. Sacks FM, Pfeffer MA, Moye LA, Rouleau JL, Rutherford JD, Cole TG, Brown L, Warnica JW, Arnold JMO, Wun CC, Davis BR, Braunwald E. The effect of pravastatin on coronary events after myocardial infarction in patients with average cholesterol levels. Cholesterol and Recurrent Events Trial Investigators. *N Engl J Med* 1996; 335(14):1001-1009.
- 70. Baseline serum cholesterol and treatment effect in the Scandinavian Simvastatin Survival Study (4S). *Lancet* 1995 May 20; 345(8960):1274-1275.

- 71. Shepherd J, Cobbe SM, Ford I, Isles CG, Lorimer AR, MacFarlane RW, McKillop JH, Packard CJ. Prevention of coronary heart disease with pravastatin in men with hypercholesterolemia. West of Scotland Coronary Prevention Study Group. *N Engl J Med* 1995; 333(20):1301-1307.
- 72. Teo KK, Yusuf S, Pfeffer M, Torp-Pedersen C, Kober L, Hall A, Pogue J, Latini R, Collins R. Effects of long-term treatment with angiotensin-converting-enzyme inhibitors in the presence or absence of aspirin: a systematic review. *Lancet* 2002 Oct 5; 360(9339):1037-1043.
- 73. Thompson AM, Hu T, Eshelbrenner CL, Reynolds K, He J, Bazzano LA. Antihypertensive treatment and secondary prevention of cardiovascular disease events among persons without hypertension: a meta-analysis. *JAMA* 2011 Mar 2; 305(9):913-922.
- 74. Wald NJ, Law MR. A strategy to reduce cardiovascular disease by more than 80%. *BMJ* 2003 Jun 28; 326(7404):1419.
- 75. Weisman SM, Graham DY. Evaluation of the benefits and risks of low-dose aspirin in the secondary prevention of cardiovascular and cerebrovascular events. *Arch Intern Med* 2002 Oct 28; 162(19):2197-2202.
- 76. Yeh RW, Sidney S, Chandra M, Sorel M, Selby JV, Go AS. Population trends in the incidence and outcomes of acute myocardial infarction. *N Engl J Med* 2010 Jun 10; 362(23):2155-2165.
- 77. Yusuf S, Sleight P, Pogue J, Bosch J, Davies R, Dagenais G. Effects of an angiotensin-converting-enzyme inhibitor, ramipril, on cardiovascular events in high-risk patients. The Heart Outcomes Prevention Evaluation Study Investigators. *N Engl J Med* 2000 Jan; 342(3):145-153.
- 78. Wong W, Jaffe M, Wong M, Dudl RJ. Implementation Study-Vohs National Quality Award. Community Implementation and Translation of Kaiser Permanente's Cardiovascular Disease Risk-Reduction Strategy. *The Permanente Journal* 2011; 15(1):36-41.
- 79. Kern LM, Ancker JS, Abramson E, Patel V, Dhopeshwarkar RV, Kaushal R. Evaluating health information technology in community-based settings: lessons learned. *J Am Med Inform Assoc* 2011 Nov; 18(6):749-753.
- 80. Rabin BA, Glasgow RE, Kerner JF, Klump MP, Brownson RC. Dissemination and implementation research on community-based cancer prevention: a systematic review. *Am J Prev Med* 2010 Apr; 38(4):443-456.
- 81. Rycroft-Malone J, Seers K, Crichton N, Chandler J, Hawkes CA, Allen C, Bullock I, Strunin L. A pragmatic cluster randomised trial evaluating three implementation interventions. *Implement Sci* 2012; 7:80.
- 82. Bero LA, Grilli R, Grimshaw JM, Harvey E, Oxman AD, Thomson MA. Closing the gap between research and practice: an overview of systematic reviews of interventions to promote the implementation of research findings. The Cochrane Effective Practice and Organization of Care Review Group. *BMJ* 1998 Aug 15; 317(7156):465-468.
- 83. Grimshaw JM, Thomas RE, MacLennan G, Fraser C, Ramsay CR, Vale L, Whitty P, Eccles MP, Matowe L, Shirran L, Wensing M, Dijkstra R, Donaldson C. Effectiveness and efficiency of guideline dissemination and implementation strategies. *Health Technol Assess* 2004 Feb; 8(6):iii-72.
- 84. Thompson DS, Estabrooks CA, Scott-Findlay S, Moore K, Wallin L. Interventions aimed at increasing research use in nursing: a systematic review. *Implement Sci* 2007; 2:15.
- 85. Hakkennes S, Dodd K. Guideline implementation in allied health professions: a systematic review of the literature. *Qual Saf Health Care* 2008 Aug; 17(4):296-300.
- 86. Schouten LM, Hulscher ME, van Everdingen JJ, Huijsman R, Grol RP. Evidence for the impact of quality improvement collaboratives: systematic review. *BMJ* 2008 Jun 28; 336(7659):1491-1494.
- 87. Godfrey CM, Harrison MB, Graham ID. A review of the use of outcome measures of evidence-based practice in guideline implementation studies in nursing, allied health professions and medicine. In: Bick D, Graham ID, eds. *Evaluating the impact of implementing evidence-based practice*. Oxford: Wiley-Blackwell, 2010, pp 189-200.
- 88. Mold JW, Aspy CA, Nagykaldi Z. Implementation of evidence-based preventive services delivery processes in primary care: an Oklahoma Physicians Resource/Research Network (OKPRN) study. *J Am Board Fam Med* 2008 Jul; 21(4):334-344.

- 89. Kolko DJ, Baumann BL, Herschell AD, Hart JA, Holden EA, Wisniewski SR. Implementation of AF-CBT by community practitioners serving child welfare and mental health: a randomized trial. *Child Maltreat* 2012 Feb; 17(1):32-46.
- 90. Soumerai SB, McLaughlin TJ, Gurwitz JH, Guadagnoli E, Hauptman PJ, Borbas C, Morris N, McLaughlin B, Gao X, Willison DJ, Asinger R, Gobel F. Effect of local medical opinion leaders on quality of care for acute myocardial infarction: a randomized controlled trial. *JAMA* 1998 May 6; 279(17):1358-1363.
- 91. Wallin L. Knowledge translation and implementation research in nursing. *Int J Nurs Stud* 2009 Apr; 46(4):576-587.
- 92. Smith JL, Williams JW, Jr., Owen RR, Rubenstein LV, Chaney E. Developing a national dissemination plan for collaborative care for depression: QUERI Series. *Implement Sci* 2008 Dec 31; 3:59. doi: 10.1186/1748-5908-3-59.:59-3.
- 93. Massoud MR, Nielson GA, Nolan K, Schall MW, Sevin C. A Framework for Spread: From Local Improvements to System-Wide Change. IHI Innovation Series white paper. Cambridge, MA: Institute for Healthcare Improvement. Available at: <a href="https://www.IHI.org">www.IHI.org</a>. Accessed on: 1-8-2013.
- 94. Paina L, Peters DH. Understanding pathways for scaling up health services through the lens of complex adaptive systems. *Health Policy Plan* 2012 Aug; 27(5):365-373.
- 95. Quanbeck AR, Gustafson DH, Ford JH, Pulvermacher A, French MT, McConnell KJ, McCarty D. Disseminating quality improvement: study protocol for a large cluster-randomized trial. *Implement Sci* 2011; 6:44.
- 96. Grimshaw J, Eccles M, Thomas R, MacLennan G, Ramsay C, Fraser C, Vale L. Toward evidence-based quality improvement. Evidence (and its limitations) of the effectiveness of guideline dissemination and implementation strategies 1966-1998. *J Gen Intern Med* 2006 Feb; 21 Suppl 2:S14-S20.
- 97. Baker J, Playle J, Nelson P, Lovell K. An evaluation of the impact of the recommendations of the Chief Nursing Officer's (England) Review of Mental Health Nursing in Mental Health Trusts and Universities in England: findings from stage one, an e-survey. *J Clin Nurs* 2010 Sep; 19(17-18):2590-2600.
- 98. US DHHS. Community Health Centers and the Affordable Care Act in 2011: Increasing Access to Affordable, Cost Effective, High Quality Care. Available at: <a href="http://www.healthcare.gov/news/factsheets/2011/08/communityhealthcenters08092011a.html">http://www.healthcare.gov/news/factsheets/2011/08/communityhealthcenters08092011a.html</a>. Accessed on: 2-20-2012.
- 99. The White House. The Obama Administration and Community Health Centers. 2012. Available at: <a href="http://www.whitehouse.gov/sites/default/files/05-01-12">http://www.whitehouse.gov/sites/default/files/05-01-12</a> community health center report.pdf. Accessed on: 06/05/2012.
- 100. Morgan D. Health centers for poor, uninsured see ranks swell. 2012. Available at: <a href="http://www.reuters.com/article/2012/05/01/us-usa-healthcare-centers-idUSBRE8401JL20120501">http://www.reuters.com/article/2012/05/01/us-usa-healthcare-centers-idUSBRE8401JL20120501</a>. Accessed on: 01/21/2013.
- 101. Lundgren L, Amodeo M, Cohen A, Chassler D, Horowitz A. Modifications of evidence-based practices in community-based addiction treatment organizations: a qualitative research study. *Addict Behav* 2011 Jun; 36(6):630-635.
- 102. Chang ET, Rose DE, Yano EM, Wells KB, Metzger ME, Post EP, Lee ML, Rubenstein LV. Determinants of Readiness for Primary Care-Mental Health Integration (PC-MHI) in the VA Health Care System. *J Gen Intern Med* 2012 Oct 5.
- 103. Gold R. The Guide to Conducting Research in the OCHIN Practice Management Data. Available at: *Kaiser Permanente Center for Health Research*.
- 104. DeVoe JE, Gold R, McIntire P, Puro J, Chauvie S, Gallia CA. Electronic health records vs Medicaid claims: completeness of diabetes preventive care data in community health centers. *Ann Fam Med* 2011 Jul; 9(4):351-358.
- 105. Gold R, DeVoe J, Shah A, Chauvie S. Insurance continuity and receipt of diabetes preventive care in a network of federally qualified health centers. *Med Care* 2009 Apr; 47(4):431-439.
- 106. Gold R, DeVoe JE, McIntire PJ, Puro JE, Chauvie SL, Shah AR. Receipt of diabetes preventive care among safety net patients associated with differing levels of insurance coverage. *J Am Board Fam Med* 2012 Jan; 25(1):42-49.

- 107. DeVoe JE, Gold R, Spofford M, Chauvie S, Muench J, Turner A, Likumahuwa S, Nelson C. Developing a network of community health centers with a common electronic health record: description of the Safety Net West Practice-based Research Network (SNW-PBRN). *J Am Board Fam Med* 2011 Sep; 24(5):597-604.
- 108. Jones B, Lightfoot A, De MM, Isler MR, Ammerman A, Nelson D, Harrison L, Motsinger B, Melvin C, Corbie-Smith G. Community-responsive research priorities: health research infrastructure. *Prog Community Health Partnersh* 2012; 6(3):339-348.
- 109. National Institutes of Health. Training Institute for Dissemination and Implementation Research in Health 2012. 2012. Available at: <a href="http://conferences.thehillgroup.com/OBSSRinstitutes/TIDIRH2012/index.html">http://conferences.thehillgroup.com/OBSSRinstitutes/TIDIRH2012/index.html</a>. Accessed on: 06/05/2012.
- 110. Cohen DJ, Balasubramanian BA, Isaacson NF, Clark EC, Etz RS, Crabtree BF. Coordination of health behavior counseling in primary care. *Ann Fam Med* 2011 Sep; 9(5):406-415.
- 111. Cohen DJ, Flocke SA, Lawson P, Casucci B. How teachable moments are co-constructed to deliver health behavior advice during primary care visits. American Academy of Communication in Health Care International Conference. South Carolina. 2007.
- 112. Cohen DJ, Crabtree BF. Evaluative criteria for qualitative research in health care: controversies and recommendations. *Ann Fam Med* 2008 Jul; 6(4):331-339.
- 113. Angier H, Gregg J, Gold R, Crocker S, Dean K, DeVoe JE. A Qualitative Assessment of Barriers and Facilitators of Access to Health Care: Oregon Family Perspectives. *In press: Academic Pediatrics* 2012.
- 114. DeVoe JE, Graham A, Krois L, Smith J, Fairbrother GL. "Mind the Gap" in children's health insurance coverage: does the length of a child's coverage gap matter? *Ambul Pediatr* 2008 Mar; 8(2):129-134.
- 115. DeVoe JE, Krois L, Edlund C, Smith J, Carlson NE. Uninsured but eligible children: are their parents insured? Recent findings from Oregon. *Med Care* 2008 Jan; 46(1):3-8.
- 116. DeVoe JE, Westfall N, Crocker S, Eigner D, Selph S, Bunce A, Wallace L. Why do some eligible families forego public insurance for their children? A qualitative analysis. *Fam Med* 2012 Jan; 44(1):39-46.
- 117. Angier H, Wiggins N, Gregg J, Gold R, DeVoe JE. Engagement of Community Health Workers In a Health Policy Research Project Through a Novel Technique: The Community Retreat Paper presented at: North American Primary Care Research Group 2011; Banff, Alberta. 2011.
- 118. Gold R, Angier H, Mangione-Smith R, Gallia C, McIntire PJ, Cowburn S, Tillotson C, DeVoe JE. Feasibility of evaluating the CHIPRA care quality measures in electronic health record data. *Pediatrics* 2012 Jul; 130(1):139-149.
- 119. Young RA, DeVoe JE. What could family income be if health insurance were more affordable? *Fam Med* 2012 Oct; 44(9):633-636.
- 120. Angier H, DeVoe JE, Tillotson CJ, Wallace LS. Changes in US Family Health Insurance Coverage Patterns: Comparing 2003 to 2008. *Family Medicine* 2013; 45(1):26-32.
- 121. Casciato A, Angier H, Milano C, Gideonse N, Gold R, DeVoe JE. A practice-based approach to demonstrate the use of pediatric quality measures in outpatient electronic health record data. *Journal of the American Board of Family Medicine* 2012; 25(5):686-693.
- 122. Saultz JW, Brown D, Stenberg S, Rdesinski RE, Tillotson CJ, Eigner D, DeVoe J. Access assured: a pilot program to finance primary care for uninsured patients using a monthly enrollment fee. *J Am Board Fam Med* 2010 May; 23(3):393-401.
- 123. Saultz JW, Heineman J, Seltzer R, Bunce A, Spires L, DeVoe J. Uninsured patient opinions about a reduced-fee retainer program at academic health center clinics. *J Am Board Fam Med* 2011 May; 24(3):304-312.
- 124. DeVoe JE, Krois L, Stenger R. Do children in rural areas still have different access to health care? Results from a statewide survey of Oregon's food stamp population. *J Rural Health* 2009; 25(1):1-7.
- 125. Young RA, DeVoe JE. Who will have health insurance in the future? An updated projection. *Ann Fam Med* 2012 Mar; 10(2):156-162.

- 126. Yamauchi M, Carlson MJ, Wright BJ, Angier H, DeVoe JE. Does Health Insurance Continuity Among Low-income Adults Impact Their Children's Insurance Coverage? *Matern Child Health J* 2012 Feb 23. [Epub ahead of print]
- 127. DeVoe JE, Tillotson CJ, Wallace LS, Lesko SE, Pandhi N. Is health insurance enough? A usual source of care may be more important to ensure a child receives preventive health counseling. *Matern Child Health J* 2012 Feb; 16(2):306-315.
- 128. DeVoe JE, Tillotson CJ, Lesko SE, Wallace LS, Angier H. The case for synergy between a usual source of care and health insurance coverage. *J Gen Intern Med* 2011 Sep; 26(9):1059-1066.
- 129. DeVoe JE, Wallace L, Selph S, Westfall N, Crocker S. Comparing type of health insurance among low-income children: a mixed methods study from Oregon. *Matern Child Health J* 2011 Nov; 15(8):1238-1248.
- 130. DeVoe JE, Tillotson CJ, Wallace LS, Angier H, Carlson MJ, Gold R. Parent and child usual source of care and children's receipt of health care services. *Ann Fam Med* 2011 Nov; 9(6):504-513.
- 131. Wallace LS, DeVoe JE, Hansen JS. Assessment of Children's Public Health Insurance Program enrollment applications: a health literacy perspective. *J Pediatr Health Care* 2011 Mar; 25(2):133-137.
- 132. Hansen JS, Wallace LS, DeVoe JE. How readable are Spanish-language Medicaid applications? *J Immigr Minor Health* 2011 Apr; 13(2):293-298.
- 133. Bauer J, Angus L, Fischler N, Rosenberg KD, Gipson TF, DeVoe J. The impact of citizenship documentation requirements on access to medicaid for pregnant women in Oregon. *Matern Child Health J* 2011 Aug; 15(6):753-758.
- 134. DeVoe JE, Ray M, Krois L, Carlson MJ. Uncertain health insurance coverage and unmet children's health care needs. *Fam Med* 2010 Feb; 42(2):121-132.
- 135. Angus L, DeVoe J. Evidence that the citizenship mandate curtailed participation in Oregon's Medicaid family planning program. *Health Aff (Millwood)* 2010 Apr; 29(4):690-698.
- 136. DeVoe JE. Educaid: what if the US systems of education and health care were more alike? *Fam Med* 2009 Oct; 41(9):652-655.
- 137. DeVoe JE, Saultz JW, Krois L, Tillotson CJ. A medical home versus temporary housing: the importance of a stable usual source of care. *Pediatrics* 2009 Nov; 124(5):1363-1371.
- 138. Wilson JM, Wallace LS, DeVoe JE. Are state Medicaid application enrollment forms readable? *J Health Care Poor Underserved* 2009 May; 20(2):423-431.
- 139. DeVoe JE, Tillotson C, Wallace LS. Uninsured children and adolescents with insured parents. *JAMA* 2008 Oct 22: 300(16):1904-1913.
- 140. DeVoe J. The unsustainable US health care system: a blueprint for change. *Ann Fam Med* 2008 May; 6(3):263-266.
- 141. DeVoe JE, Petering R, Krois L. A usual source of care: supplement or substitute for health insurance among low-income children? *Med Care* 2008 Oct; 46(10):1041-1048.
- 142. Carlson MJ, DeVoe J, Wright BJ. Short-term impacts of coverage loss in a Medicaid population: early results from a prospective cohort study of the Oregon Health Plan. *Ann Fam Med* 2006 Sep; 4(5):391-398.
- 143. DeVoe J, Krois L. Issue Brief: Covering Kids, Children's Access to Healthcare. Salem, OR: Office for Oregon Health Policy and Research. Available at: <a href="http://www.oregon.gov/oha/OHPR/RSCH/docs/ckidsbrief\_final.pdf">http://www.oregon.gov/oha/OHPR/RSCH/docs/ckidsbrief\_final.pdf</a>. Accessed on: 1-10-2013.
- 144. Wright BJ, Carlson MJ, Edlund T, DeVoe J, Gallia C, Smith J. The impact of increased cost sharing on Medicaid enrollees. *Health Aff (Millwood)* 2005 Jul; 24(4):1106-1116.
- 145. Who will have health insurance in 2025? Am Fam Physician 2005 Nov 15; 72(10):1989.
- 146. DeVoe J, Smith J, Edlund C, Krois L. Issue Brief: Employer-Sponsored Private Health Insurance Costs, 1997-2002. 2005.

- 147. Solotaroff R, DeVoe J, Wright BJ, Smiths J, Boone J, Edlund T, Carlson MJ. Medicaid programme changes and the chronically ill: early results from a prospective cohort study of the Oregon Health Plan. *Chronic Illn* 2005 Sep; 1(3):191-205.
- 148. DeVoe JE, Wallace LS, Pandhi N, Solotaroff R, Fryer GE, Jr. Comprehending care in a medical home: a usual source of care and patient perceptions about healthcare communication. *J Am Board Fam Med* 2008 Sep; 21(5):441-450.
- 149. DeVoe JE, Fryer GE, Phillips R, Green L. Receipt of preventive care among adults: insurance status and usual source of care. *Am J Public Health* 2003 May; 93(5):786-791.
- 150. DeVoe J. A policy transformed by politics: the case of the 1973 Australian Community Health Program. *J Health Polit Policy Law* 2003 Feb; 28(1):77-108.
- 151. De Voe JE, Short SD. A shift in the historical trajectory of medical dominance: the case of Medibank and the Australian doctors' lobby. *Soc Sci Med* 2003 Jul; 57(2):343-353.
- 152. Tilden VP, Nelson CA, Dunn PM, Donius M, Tolle SW. Nursing's perspective on improving communication about nursing home residents' preferences for medical treatments at end of life. *Nurs Outlook* 2000 May; 48(3):109-115.
- 153. Tilden VP, Tolle SW, Nelson CA, Fields J. Family decision-making to withdraw life-sustaining treatments from hospitalized patients. *Nurs Res* 2001 Mar; 50(2):105-115.
- 154. Norton SA, Tilden VP, Tolle SW, Nelson CA, Eggman ST. Life support withdrawal: communication and conflict. *Am J Crit Care* 2003 Nov; 12(6):548-555.
- 155. Hickman SE, Nelson CA, Moss AH, Hammes BJ, Terwilliger A, Jackson A, Tolle SW. Use of the Physician Orders for Life-Sustaining Treatment (POLST) paradigm program in the hospice setting. *J Palliat Med* 2009 Feb; 12(2):133-141.
- 156. Hickman SE, Nelson CA, Perrin NA, Moss AH, Hammes BJ, Tolle SW. A comparison of methods to communicate treatment preferences in nursing facilities: traditional practices versus the physician orders for life-sustaining treatment program. *J Am Geriatr Soc* 2010 Jul; 58(7):1241-1248.
- 157. Hickman SE, Nelson CA, Moss AH, Tolle SW, Perrin NA, Hammes BJ. The consistency between treatments provided to nursing facility residents and orders on the physician orders for life-sustaining treatment form. *J Am Geriatr Soc* 2011 Nov; 59(11):2091-2099.
- 158. DeVoe JE, Likumahuwa S, Eiff MP, Nelson CA, Carroll JE, Hill CN, Gold R, Kullberg PA. Lessons learned and challenges ahead: report from the OCHIN Safety Net West practice-based research network (PBRN). *J Am Board Fam Med* 2012 Sep; 25(5):560-564.
- 159. Hickman SE, Cartwright JC, Nelson CA, Knafl K. Compassion and vigilance: investigators' strategies to manage ethical concerns in palliative and end-of-life research. *J Palliat Med* 2012 Aug; 15(8):880-889.
- 160. Brody KK, Perrin N. Advanced illness index: Identifying vulnerable persons with complex care needs. (submitted)
- 161. Brown JB, Nichols GA, Bachman K, DeBar L, Moiel D, Perrin N. Medical care costs before and after Bariatric surgery. *Obes Res* 2004;12:A149
- 162. Feldstein AC, Perrin NA, Unitan R, Rosales AG, Nichols GA, Smith DH, Schneider J, Davino CM, Zhou YY, Lee NL. Effect of a patient panel-support tool on care delivery. *Am J Manag Care* 2010 Oct 1; 16(10):e256-e266.
- 163. Feldstein AC, Smith DH, Perrin N, Yang X, Simon SR, Krall M, Sittig DF, Ditmer D, Platt R, Soumerai SB. Reducing warfarin medication interactions: an interrupted time series evaluation. *Arch Intern Med* 2006 May 8; 166(9):1009-1015.
- 164. Feldstein AC, Perrin N, Liles EG, Smith DH, Rosales AG, Schneider JL, Lafata JE, Myers RE, Mosen DM, Glasgow RE. Primary care colorectal cancer screening recommendation patterns: associated factors and screening outcomes. *Med Decis Making* 2012 Jan; 32(1):198-208.
- 165. Feldstein AC, Nichols GA, Smith DH, Stevens VJ, Bachman K, Rosales AG, Perrin N. Weight change in diabetes and glycemic and blood pressure control. *Diabetes Care* 2008 Oct; 31(10):1960-1965.

- 166. Feldstein AC, Nichols GA, Smith DH, Rosales AG, Perrin N. Weight change and glycemic control after diagnosis of type 2 diabetes. *J Gen Intern Med* 2008 Jun; epub ahead of print.
- 167. Simon SR, Smith DH, Feldstein AC, Perrin N, Yang X, Zhou Y, Platt R, Soumerai SB. Computerized prescribing alerts and group academic detailing to reduce the use of potentially inappropriate medications in older people. *J Am Geriatr Soc* 2006 Jun; 54(6):963-968.
- 168. Smith DH, Feldstein AC, Perrin NA, Yang X, Rix MM, Raebel MA, Magid DJ, Simon SR, Soumerai SB. Improving laboratory monitoring of medications: an economic analysis alongside a clinical trial. *Am J Manag Care* 2009 May; 15(5):281-289.
- Ash JS, Sittig DF, Wright A, McMullen C, Shapiro M, Bunce A, Middleton B. Clinical decision support in small community practice settings: a case study. *J Am Med Inform Assoc* 2011 Nov; 18(6):879-882.
- 170. McMullen CK, Ash JS, Sittig DF, Bunce A, Guappone K, Dykstra R, Carpenter J, Richardson J, Wright A. Rapid assessment of clinical information systems in the healthcare setting: an efficient method for time-pressed evaluation. *Methods Inf Med* 2011; 50(4):299-307.
- 171. Ash JS, Sittig DF, Guappone KP, Dykstra RH, Richardson J, Wright A, Carpenter J, McMullen C, Shapiro M, Bunce A, Middleton B. Recommended practices for computerized clinical decision support and knowledge management in community settings: a qualitative study. *BMC Med Inform Decis Mak* 2012; 12:6.
- 172. Ash JS, Sittig DF, McMullen C, McCormack J, Wright A, Bunce A, Wasserman J, Mohan V, Cohen D, Shapiro M, Middleton B. Studying the Vendor Perspective on Clinical Decision Support. American Medical Informatics Association Annual Symposium Proceedings 2011, OHSU, Portland, OR. 2011.
- 173. Abramson E, Patel V, Malhotra S, Pfoh E, Osorio S, Cheriff A, Cole C, Bunce A, Ash JS, Kaushal R. Physician experiences transitioning between an older versus newer electronic health record for electronic prescribing. *International Journal of Medical Informatics* 2012 Aug; 81(8):539-548.
- 174. Chen ES, Melton GB, Burdick TE, Rosenau PT, Sarkar IN. Characterizing the use and contents of free-text family history comments in the electronic health record. *AMIA Annu Symp Proc* 2012; 2012:85-92.
- 175. Deyo RA, Smith DH, Johnson ES, Donovan M, Tillotson CJ, Yang X, Petrik AF, Dobscha SK. Opioids for back pain patients: primary care prescribing patterns and use of services. *J Am Board Fam Med* 2011 Nov; 24(6):717-727.
- 176. Smith DH, Johnson ES, Thorp ML, Yang X, Petrik A, Platt RW, Crispell K. Predicting poor outcomes in heart failure. *Perm J* 2011; 15(4):4-11.
- 177. Smith DH, Raebel MA, Chan KA, Johnson ES, Petrik AF, Weiss JR, Yang X, Feldstein A. An economic evaluation of a laboratory monitoring program for renin-angiotensin system agents. *Med Decis Making* 2011 Mar; 31(2):315-324.
- 178. Smith DH, Johnson ES, Thorp ML, Yang X, Neil N. Hyperparathyroidism in chronic kidney disease: a retrospective cohort study of costs and outcomes. *J Bone Miner Metab* 2009; 27(3):287-294.
- 179. Ogawa H, Nakayama M, Morimoto T, Uemura S, Kanauchi M, Doi N, Jinnouchi H, Sugiyama S, Saito Y. Low-dose aspirin for primary prevention of atherosclerotic events in patients with type 2 diabetes: a randomized controlled trial. *JAMA* 2008 Nov 12; 300(18):2134-2141.
- Belch J, MacCuish A, Campbell I, Cobbe S, Taylor R, Prescott R, Lee R, Bancroft J, MacEwan S, Shepherd J, Macfarlane P, Morris A, Jung R, Kelly C, Connacher A, Peden N, Jamieson A, Matthews D, Leese G, McKnight J, O'Brien I, Semple C, Petrie J, Gordon D, Pringle S, MacWalter R. The prevention of progression of arterial disease and diabetes (POPADAD) trial: factorial randomised placebo controlled trial of aspirin and antioxidants in patients with diabetes and asymptomatic peripheral arterial disease. BMJ 2008 Oct 16; 337:a1840. doi: 10.1136/bmj.a1840.:a1840.
- 181. Colhoun HM, Betteridge DJ, Durrington PN, Hitman GA, Neil HAW, Livingstone SJ, Thomason MJ, Mackness MI, Charlton-Menys V, Fuller JH, on behalf of the CARDS investigators. Primary prevention of cardiovascular disease with atorvastatin in type 2 diabetes in the Collaborative Atorvastatin Diabetes Study (CARDS): multicentre randomised placebo-controlled trial. *Lancet* 2004 Aug 21; 364:685-696.
- 182. Kearney PM, Blackwell L, Collins R, Keech A, Simes J, Peto R, Armitage J, Baigent C. Efficacy of cholesterol-lowering therapy in 18,686 people with diabetes in 14 randomised trials of statins: a meta-analysis. *Lancet* 2008 Jan 12; 371(9607):117-125.

- 183. Lewis EJ, Hunsicker LG, Bain RP, Rohde RD. The effect of angiotensin-converting-enzyme inhibition on diabetic nephropathy. *New England Journal of Medicine* 1993; 329(20):1456-1462.
- 184. Hansson L, Zanchetti A, Carruthers SG, Dahlof B, Elmfeldt D, Julius S, Menard J, Rahn KH, Wedel H, Westerling S. Effects of intensive blood pressure lowering and low dose aspirin in patients with hypertension: principle results of the Hypertension Optimal Treatment (HOT) randomised trial. HOT Study Group. *Lancet* 1998; 351:1755-1762.
- 185. Hayden M, Pignone M, Phillips C, Mulrow C. Aspirin for the primary prevention of cardiovascular events: a summary of the evidence for the U.S. Preventive Services Task Force. *Ann Intern Med* 2002 Jan 15; 136(2):161-172.
- 186. Antiplatelet Trialists Collaborative. Collaborative overview of randomised trials of antiplatelet therapy, I: Prevention of death, myocardial infarction, and stroke by prolonged antiplatelet therapy in various categories of patients. *BMJ* 1994; 308:81-106.
- 187. UK Prospective Diabetes Study Group. Efficacy of atenolol and captopril in reducing risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 39. *BMJ* 1998 Sep 12; 317(7160):713-720.
- 188. UK Prospective Diabetes Study Group. Tight blood pressure control and risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 38. *BMJ* 1998 Sep 12; 317(7160):703-713.
- 189. American Diabetes Association. Standards of Medical Care in Diabetes--2008. *Diabetes Care* 2008 Jan; 31(Supp 1):S12-S54.
- 190. Pettay HS, Branthaver B, Cristobal K, Wong M. The care management institute: harvesting innovation, maximizing transfer. *Perm J* 2005; 9(4):37-39.
- 191. Community Clinics Health Network. Community Clinics Health Network. Community Clinics Health Network Final Report to Kaiser Permanente. Implementation of the Aspirin, Lisinopril, Lovastatin (A.L.L.) Intervention in Community Clinics Project Period: December 1, 2005 to December 1, 2007. 2008.
- 192. Jilcott S, Ammerman A, Sommers J, Glasgow RE. Applying the RE-AIM framework to assess the public health impact of policy change. *Ann Behav Med* 2007 Oct; 34(2):105-114.
- 193. Crabtree BF, Miller WL, Stange KC. Understanding practice from the ground up. *J Fam Pract* 2001 Oct; 50(10):881-887.
- 194. Crabtree BF, Miller WL, Aita VA, Flocke SA, Stange KC. Primary care practice organization and preventive services delivery: a qualitative analysis. *J Fam Pract* 1998 May; 46(5):403-409.
- 195. Miller WL, McDaniel RR, Jr., Crabtree BF, Stange KC. Practice jazz: understanding variation in family practices using complexity science. *J Fam Pract* 2001 Oct; 50(10):872-878.
- 196. Miller WL, Crabtree BF, McDaniel R, Stange KC. Understanding change in primary care practice using complexity theory. *J Fam Pract* 1998 May; 46(5):369-376.
- 197. Balasubramanian BA, Chase SM, Nutting PA, Cohen DJ, Strickland PA, Crosson JC, Miller WL, Crabtree BF. Using Learning Teams for Reflective Adaptation (ULTRA): insights from a team-based change management strategy in primary care. *Ann Fam Med* 2010 Sep; 8(5):425-432.
- 198. Lukas CV, Meterko MM, Mohr D, Seibert MN, Parlier R, Levesque O, Petzel RA. Implementation of a clinical innovation: the case of advanced clinic access in the Department of Veterans Affairs. *J Ambul Care Manage* 2008 Apr; 31(2):94-108.
- 199. Solberg LI. Improving medical practice: a conceptual framework. Ann Fam Med 2007 May; 5(3):251-256.
- 200. Subramanian S, Naimoli J, Matsubayashi T, Peters DH. Do we have the right models for scaling up health services to achieve the Millennium Development Goals? *BMC Health Serv Res* 2011; 11:336.
- 201. Janovsky K, Peters DH, Arur A, Sundaram S. Improving health services and strengthening health systems: adopting and implementing innovative strategies. Making Health Systems Work, Working Paper No. 5. Geneva: World Health Organization, Evidence and Information for Policy. 2006.
- 202. Taylor EF, Machta RM, Meyers DS, Genevro J, Peikes DN. Enhancing the primary care team to provide redesigned care: the roles of practice facilitators and care managers. *Ann Fam Med* 2013 Jan; 11(1):80-83.

- 203. Munoz M, Pronovost P, Dintzis J, Kemmerer T, Wang NY, Chang YT, Efird L, Berenholtz SM, Golden SH. Implementing and evaluating a multicomponent inpatient diabetes management program: putting research into practice. *Jt Comm J Qual Patient Saf* 2012 May; 38(5):195-206.
- 204. Weir C, McLeskey N, Brunker C, Brooks D, Supiano MA. The role of information technology in translating educational interventions into practice: an analysis using the PRECEDE/PROCEED model. *J Am Med Inform Assoc* 2011 Nov; 18(6):827-834.
- 205. Helfrich CD, Damschroder LJ, Hagedorn HJ, Daggett GS, Sahay A, Ritchie M, Damush T, Guihan M, Ullrich PM, Stetler CB. A critical synthesis of literature on the promoting action on research implementation in health services (PARIHS) framework. *Implement Sci* 2010 Oct 25; 5:82. doi: 10.1186/1748-5908-5-82.:82-85.
- 206. Simpson DD, Dansereau DF. Assessing organizational functioning as a step toward innovation. *Sci Pract Perspect* 2007 Apr; 3(2):20-28.
- 207. Jaen CR, Crabtree BF, Palmer RF, Ferrer RL, Nutting PA, Miller WL, Stewart EE, Wood R, Davila M, Stange KC. Methods for evaluating practice change toward a patient-centered medical home. *Ann Fam Med* 2010; 8 Suppl 1:S9-20.
- 208. Simon JS, Rundall TG, Shortell SM. Adoption of order entry with decision support for chronic care by physician organizations. *J Am Med Inform Assoc* 2007 Jul; 14(4):432-439.
- 209. Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: Development and validation. *Journal of Chronic Disease* 1987; 40(5):373-383.
- 210. de Groot V, Beckerman H, Lankhorst GJ, Bouter LM. How to measure comorbidity. a critical review of available methods. *J Clin Epidemiol* 2003 Mar; 56(3):221-229.
- 211. Fleuren M, Wiefferink K, Paulussen T. Determinants of innovation within health care organizations: literature review and Delphi study. *Int J Qual Health Care* 2004 Apr; 16(2):107-123.
- 212. Daley CM, James AS, Filippi M, Weir M, Braiuca S, Kaur B, Choi WS, Greiner KA. American Indian Community Leader and Provider Views of Needs and Barriers to Colorectal Cancer Screening. *J Health Dispar Res Pract* 2012; 5(2).
- 213. Ratanawongsa N, Crosson JC, Schillinger D, Karter AJ, Saha CK, Marrero DG. Getting under the skin of clinical inertia in insulin initiation: the Translating Research Into Action for Diabetes (TRIAD) Insulin Starts Project. *Diabetes Educ* 2012 Jan; 38(1):94-100.
- 214. Stamatakis KA, McQueen A, Filler C, Boland E, Dreisinger M, Brownson RC, Luke DA. Measurement properties of a novel survey to assess stages of organizational readiness for evidence-based interventions in community chronic disease prevention settings. *Implement Sci* 2012 Jul 16; 7:65. doi: 10.1186/1748-5908-7-65.:65-67.
- 215. Solberg LI, Asche SE, Margolis KL, Whitebird RR. Measuring an organization's ability to manage change: the change process capability questionnaire and its use for improving depression care. *Am J Med Qual* 2008 May; 23(3):193-200.
- Emmons KM, Weiner B, Fernandez ME, Tu SP. Systems antecedents for dissemination and implementation: a review and analysis of measures. *Health Educ Behav* 2012 Feb; 39(1):87-105.
- 217. Cohen DJ, Tallia AF, Crabtree BF, Young DM. Implementing health behavior change in primary care: lessons from prescription for health. *Ann Fam Med* 2005 Jul; 3 Suppl 2:S12-S19.
- 218. Cohen DJ, Crabtree BF, Etz RS, Balasubramanian BA, Donahue KE, Leviton LC, Clark EC, Isaacson NF, Stange KC, Green LW. Fidelity versus flexibility: translating evidence-based research into practice. *Am J Prev Med* 2008 Nov; 35(5 Suppl):S381-S389.
- 219. Etz RS, Cohen DJ, Woolf SH, Holtrop JS, Donahue KE, Isaacson NF, Stange KC, Ferrer RL, Olson AL. Bridging primary care practices and communities to promote healthy behaviors. *Am J Prev Med* 2008 Nov; 35(5 Suppl):S390-S397.
- 220. Cohen DJ, Leviton LC, Isaacson NF, Tallia AF, Crabtree BF. Online diaries for qualitative evaluation : Gaining real-time insights. *Am J Evaluation* 2006;(27):163.
- 221. Patton M. Qualitative Evaluation and Research Methods. Thousand Oaks, CA: Sage; 2002.

- 222. Argyris C, Schon D. Theory in Practice. San Francisco: Jossey-Bass; 1974.
- 223. Denzin N, Lincoln Y. *The Sage Handbook of Qualitative Research (4th ed)*. Thousand Oaks, CA: Sage; 2011.
- 224. Beebe J. Rapid Assessment Process: An Introduction. Walnut Creek, CA: AltaMira Press; 2001.
- 225. Bernard H. Research methods in anthropology: Qualitative and quantitative approaches. Thousand Oaks, CA: Sage; 1994.
- 226. Crabtree BF, Miller WL. Doing qualitative research. Newbury Park, CA: Sage; 1992.
- 227. Wagner AK, Soumerai SB, Zhang F, Ross-Degnan D. Segmented regression analysis of interrupted time series studies in medication use research. *J Clin Pharm Ther* 2002 Aug; 27(4):299-309.
- 228. Gillings D, Makuc D, Siegel E. Analysis of interrupted time series mortality trends: an example to evaluate regionalized perinatal care. *Am J Public Health* 1981 Jan: 71(1):38-46.
- 229. Gold R, Whitlock EP, Patnode CD, McGinnis PS, Buckley DI, Morris C. Prioritizing research needs based on a systematic evidence review: a pilot process for engaging stakeholders. *Health Expect* 2011 Aug 12; doi: 10.1111/j.1369-7625.2011.00716.x. [Epub ahead of print].
- 230. DeVoe JE, Wallace LS, Fryer GE, Jr. Measuring patients' perceptions of communication with healthcare providers: do differences in demographic and socioeconomic characteristics matter? *Health Expect* 2009 Mar; 12(1):70-80.
- 231. Bunce A, Guest G, Searing H, Frajzyngier V, Riwa P, Kanama J, Achwal I. Factors affecting vasectomy acceptability in Tanzania. *Int Fam Plan Perspect* 2007 Mar; 33(1):13-21.
- 232. Guest G, Bunce A, Johnson L. How Many Interviews Are Enough? An Experiment with Data Saturation and Variability. *Field Methods* 2006 Feb; 18(1):59-82.
- Cohen D, DiCicco-Bloom B, Strickland PO, Headley A, Orzano J, Levine J, Scott J, Crabtree B.
   Opportunistic approaches for delivering preventive care in illness visits. *Prev Med* 2004 May; 38(5):565-573.
- 234. Balasubramanian BA, Cohen DJ, Clark EC, Isaacson NF, Hung DY, Dickinson LM, Fernald DH, Green LA, Crabtree BF. Practice-level approaches for behavioral counseling and patient health behaviors. *Am J Prev Med* 2008 Nov; 35(5 Suppl):S407-S413.
- 235. Hung DY, Glasgow RE, Dickinson LM, Froshaug DB, Fernald DH, Balasubramanian BA, Green LA. The chronic care model and relationships to patient health status and health-related quality of life. *Am J Prev Med* 2008 Nov; 35(5 Suppl):S398-S406.
- 236. Orzano AJ, Cohen D, Scott JG, Crabtree BF. Closing the vaccine gap among toddlers in N.J. family physicians' practices. *J Okla State Med Assoc* 2005 Sep; 98(9):438-442.
- 237. Scott JG, Cohen D, DiCicco-Bloom B, Miller WL, Stange KC, Crabtree BF. Understanding healing relationships in primary care. *Ann Fam Med* 2008 Jul; 6(4):315-322.
- 238. Scott JG, Cohen D, DiCicco-Bloom B, Orzano AJ, Gregory P, Flocke SA, Maxwell L, Crabtree B. Speaking of weight: how patients and primary care clinicians initiate weight loss counseling. *Prev Med* 2004 Jun; 38(6):819-827.
- 239. Scott JG, Cohen D, DiCicco-Bloom B, Orzano AJ, Jaen CR, Crabtree BF. Antibiotic use in acute respiratory infections and the ways patients pressure physicians for a prescription. *J Fam Pract* 2001 Oct; 50(10):853-858.
- 240. Lincoln Y, Guba EG. Naturalistic inquiry. Newberry Park, CA: Sage; 1985.
- 241. Berg BL. Qualitative Research Methods for the Social Sciences, 7<sup>th</sup> ed. Boston: Allyn and Bacon; 2009.
- 242. Spradley JP. *The Ethnographic Interview*. New York: Rinehart and Winston; 1979.
- 243. Glaser BG, Strauss AL. *The Discovery of Grounded Theory: Strategies for Qualitative Research.* New York: Sociology Press; 1967.
- 244. Strauss A, Corbin J. Basics of qualitative research: Techniques and procedures for developing grounded theory (2<sup>nd</sup> ed.). Thousand Oaks, CA: Sage; 1998.

- 245. Charmaz K. Grounded Theory Methods in Social Justice Research. In: Denzin NK, Lincoln YS, eds. *The SAGE Handbook of Qualitative Research, 4<sup>th</sup> ed.* Thousand Oaks, CA: Sage Publications, Inc., 2011, pp 359-380.
- 246. Borkan J. Immersion/crystallization. In: Crabtree BF, Miller WL, eds. *Doing qualitative research.* Thousand Oaks, CA: Sage Publications, Inc., 1999, pp 179-194.
- 247. Miller WL, Crabtree BF. *The dance of interpretation. Doing Qualitative Research, 2nd Ed.* Thousand Oaks, CA: Sage Publications, Inc.; 1999.
- 248. Crabtree BF, Miller WL. *Doing Qualitative Research, 2nd Ed.* Thousand Oaks, CA: Sage Publications, Inc.; 1999.
- 249. Teddlie C, Tashakkori A. Mixed Methods Research: Contemporary Issues in an Emerging Field. In: Denzin N, Lincoln Y, eds. *The SAGE Handbook of Qualitative Research*, 4<sup>th</sup> ed.2011, pp 285-299.
- 250. Aarons GA, Green AE, Palinkas LA, Self-Brown S, Whitaker DJ, Lutzker JR, Silovsky JF, Hecht DB, Chaffin MJ. Dynamic adaptation process to implement an evidence-based child maltreatment intervention. *Implement Sci* 2012; 7:32.
- 251. Creswell J, Plano Clark V. *Designing and Conducting Mixed Methods Research*. Thousand Oaks, CA: Sage; 2007.
- 252. Tashakkori A, Teddlie C. *Handbook of Mixed Methods in Social & Behavioral Research*. Thousand Oaks: Sage; 2003.
- 253. Crabtree BF, Chase SM, Wise CG, Schiff GD, Schmidt LA, Goyzueta JR, Malouin RA, Payne SM, Quinn MT, Nutting PA, Miller WL, Jaen CR. Evaluation of patient centered medical home practice transformation initiatives. *Med Care* 2011 Jan; 49(1):10-16.
- 254. Mullins CD, Whicher D, Reese ES, Tunis S. Generating evidence for comparative effectiveness research using more pragmatic randomized controlled trials. *Pharmacoeconomics* 2010; 28(10):969-976.
- 255. Norris S, Atkins D, Bruening W, Fox S, Johnson E, Kane R, Morton SC, Oremus M, Ospina M, Randhawa G, Schoelles K, Shekelle P, Viswanathan M. Selecting observational studies for comparing medical interventions. In: Agency for Healthcare Research and Quality. Methods Guide for Comparative Effectiveness Reviews [posted June 2010]. Rockville, MD. Available at: <a href="http://effectivehealthcare.ahrq.gov/ehc/products/196/454/MethodsGuideNorris">http://effectivehealthcare.ahrq.gov/ehc/products/196/454/MethodsGuideNorris</a> 06042010.pdf. Accessed on: 1-28-2013.
- 256. Desai JR, Wu P, Nichols GA, Lieu TA, O'Connor PJ. Diabetes and asthma case identification, validation, and representativeness when using electronic health data to construct registries for comparative effectiveness and epidemiologic research. *Med Care* 2012 Jul; 50 Suppl:S30-S35.

